CLINICAL TRIAL: NCT06343545
Title: The Impact of a Multicomponent Telemedicine-Based Intervention on Quality of Life in Adults With Respiratory Failure Requiring Mechanical Ventilation: a Cluster Stepped-Wedge Randomized Clinical Trial (Tele-Rehab MV Trial)
Brief Title: Evaluation of the Impact of Telerehabilitation Strategies and Early Discharge After Respiratory Failure
Acronym: Rehab
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Rehab_PROADI
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Acute Respiratory Failure
Keywords: acute respiratory failure; rehabilitation; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care; Rehabilitation

STUDY DESIGN:
Intervention Model Description: Cluster crossover randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Other): Standard of care provided by participating hospitals
  Interventions: Behavioral: Standard of Care
- Rehabilitation (Experimental): An implementation bundle of measures to improve outcomes in intensive care unit, hospital, and after hospital discharge, including rehabilitation at home performed through telemedicine.
  Interventions: Behavioral: Standard of Care; Behavioral: Rehabilitation

INTERVENTIONS:
Behavioral: Standard of Care — Standard of Care provided by enrolling hospitals
Behavioral: Rehabilitation — An implementation bundle of measures to improve outcomes in intensive care unit, hospital, and after hospital discharge, including rehabilitation at home performed through telemedicine.
  Arms: Rehabilitation

SUMMARY:
To evaluate, through a randomized clinical trial in groups/clusters (stepped wedge), the impact of specific bundles for disability prevention and early rehabilitation, focused on 3 domains (ICU, Ward and post-discharge), on health-related quality of life and other long- and short-term outcomes in critically ill patients affected by hypoxemic acute respiratory failure with suspected COVID-19.

DETAILED DESCRIPTION:
Patients with severe forms of hypoxemic acute respiratory failure have persistent symptoms after hospital discharge, which seem to be mediated mainly by the need for mechanical ventilation. One of the main etiologies of hypoxemic acute respiratory failure is still COVID-19 in its endemic form. According to the World Health Organization (WHO), approximately 10 to 20% of people affected by COVID-19 develop persistent symptoms (lasting more than 3 months) in a condition described as Long COVID [1]. These symptoms can affect multiple organ systems (including respiratory, cardiovascular, musculoskeletal and nervous systems) and health domains (physical and mental domains, for example). A systematic review identified more than 50 symptoms potentially associated with Long COVID, including fatigue, muscle weakness, cough, dyspnea, difficulty concentrating, anosmia, headache, joint pain, insomnia, and anxiety were the most frequently reported. Such findings are similar in broader populations, including those with other forms of hypoxemic acute respiratory failure.

Observational studies demonstrate a consistent association between Long COVID and negative impacts on functionality, quality of life, hospitalizations, and costs. Two cohort studies conducted in the United States with COVID-19 hospitalization survivors (whose sum totals more than 2700 participants) found 60-day rehospitalization rates greater than 15%. Notably, about 48% of participants in one of these studies were financially distressed by COVID-19.

Although the occurrence of prolonged post-COVID symptoms does not depend exclusively on the severity of the initial SARS-CoV-2 infection, patients who require hospitalization for severe acute COVID-19 are those who have a higher prevalence of Long COVID and intensity of disabilities. In a study of more than 1700 COVID-19 survivors in China, more severe COVID-19 cases were associated with a higher risk of persistent symptoms, reduced physical capacity, muscle weakness, reduced ability to diffuse carbon monoxide (a test that evaluates the oxygenation capacity of the lungs), and an impact on quality of life. In this population of severe cases, it is believed that the prolonged effects of SARS-CoV-2 infection are added to the physical, cognitive, and mental health sequelae typically associated with critical illness (resulting from organ dysfunctions and intensive treatments, for example), potentiating the impact on the long-term health of COVID-19 survivors.

In scenarios similar to those of severe COVID-19, such as sepsis and acute respiratory distress syndrome, the implementation of mechanical ventilation release bundles, screening and early rehabilitation while still in the hospital ward, the adequate transmission of continuity of care to primary care, and the provision of access to rehabilitation after hospital discharge have shown the potential to accelerate the recovery of people affected by sequelae related to critical illnesses. However, these findings are based on preliminary studies that do not confirm their benefit in a large sample and with adequate methodology. In the broadest sense, the early initiation of interventions is an essential aspect to improve outcomes. When added to the delay in defining the etiology of the hypoxemic acute respiratory condition, it is imperative that the measures be applied in an equitable manner in the case of suspected COVID-19 and maintained even if the final diagnosis is not COVID-19. It would be ethically questionable to withdraw a potentially beneficial intervention from an at-risk population merely because it is not COVID-19, given the immense impact of acute respiratory failure on long-term quality of life.

Given the current scenario in Brazil, with more than 36 million people with a history of SARS-CoV-2 infection, it is estimated that more than 1 million people have been affected by Long COVID. Given this magnitude of cases, it is likely that during the coming years, due to the sequelae of COVID-19, the demand on the Unified Health System (SUS) for physical and mental rehabilitation services will increase. In this imminent situation, it is essential to investigate effective and pragmatic strategies, such as those described above, aimed at preventing and rehabilitating sequelae related to Long COVID, especially in patients affected by severe forms of COVID-19. Thus, a randomized clinical trial, the gold standard for evaluating interventions, will have the potential to support public policies for post-COVID-19 rehabilitation with accurate and generalizable information to the Brazilian context. The inclusion of patients with a suspected, but not confirmed, condition will allow a greater generalization of the results and early initiation of intervention in patients with other equally relevant pathologies with similar potential benefits.

Therefore, we propose a process improvement implementation study, with a design based on the allocation of hospitals (clusters) in a sequential manner (stepped wedge), to evaluate whether the implementation of care bundles in intensive care units, wards and post-discharge is capable of improving the quality of life in patients admitted to the ICU with hypoxemic acute respiratory failure within 90 days after discharge hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 18 years
2. Need for ICU admission due to hypoxemic acute respiratory failure with suspected COVID-19
3. Need for invasive mechanical ventilation.

Exclusion Criteria:

1. Severe underlying disease with a life expectancy of less than 3 months;
2. Absence of a responsible family member for cases of patients with communication difficulties (aphasia, severe cognitive impairment, non-native speakers of Portuguese);
3. Absence of telephone contact;
4. Participants already included in the study;
5. Unavailability to carry out telephone follow-ups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-10-14 (Estimated); Study Completion 2025-10-14 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 90 days after hospital discharge
  Health-related quality of life assessed by the Brazilian version of the 5-dimension, 3-level EuroQol scale (EQ-5D-3L)

SECONDARY OUTCOMES:
Mortality | 90 days
  All cause mortality
Days alive and free of hospital | 90 days since intensive care unit admission
  Days alive and free of hospital (not hospitalized)
Rehospitalization | 30 days after hospital discharge
  New hospitalization
Return to work | 90 days after hospital discharge
  Return to work or usual activities (work, study)
Anxiety and Depression | 90 days
  Anxiety and depression measured according to Hospital Anxiety and Depression Scale
New disability | 90 days
  Incidence of new disabilities for instrumental activities of daily living assessed by the Lawton & Brody scale
Disability | 90 days
  Prevalence of moderate, severe, or total physical disability assessed by the modified Barthel Index
Clinical Status | 90 days
  Ordinal scale from using World Health Organization
Cognitive impairment | 90 days
  Prevalence of cognitive impairment assessed by the Telephone Interview for Cognitive Status

CONTACTS AND LOCATIONS:
Overall Officials: Adriano Pereira, Study Chair — Hospital Israelita Albert Einstein
Locations (20):
- Brazil (20):
  - Hospital de Emergência Dr. Daniel Houly, Arapiraca, Alagoas
  - Fundação de Medicina Tropical Dr. Heitor Vieira Dourado, Manaus, Amazonas
  - Hospital de Messejana Dr. Carlos Alberto Studart Gomes (HM), Fortaleza, Ceará
  - Hospital Regional Norte - HRN, Sobral, Ceará
  - Hospital Municipal de Salvador, Salvador, Estado de Bahia
  - Hospital Geral de Vitória da Conquista, Vitória da Conquista, Estado de Bahia
  - Hospital Regional de Samambaia, Brasília, Federal District
  - Hospital Municipal Aparecida de Goiania - HMAP, Aparecida de Goiânia, Goiás
  - Hospital Estadual de Doenças Tropicais Dr. Anuar Auad, Goiânia, Goiás
  - Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Hospital Universitário - Universidade Estadual de Londrina, Londrina, Paraná
  - Hospital Municipal Pedro I, Campina Grande, Paraíba
  - Instituto de Medicina Integral "Prof. Fernando Figueira" - IMIP, Recife, Pernambuco
  - Hospital Estadual Dirceu Arcoverde, Parnaíba, Piauí
  - Hospital Municipal Ronaldo Gazolla, Rio de Janeiro, Rio de Janeiro
  - Hospital São Sebastião Martir, Venâncio Aires, Rio Grande do Sul
  - Centro De Pesquisa Em Medicina Tropical - CEPEM, Porto Velho, Rondônia
  - Hospital Geral de Roraima - HGR, Boa Vista, Roraima
  - Hospital Geral e Maternidade Tereza Ramos, Lages, Santa Catarina
  - Hospital Regional de Augustinópolis, Augustinópolis, Tocantins

IPD SHARING:
Plan to Share IPD: Yes
Data belongs to Brazilian Ministry of Health. May be shared upon agreement
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Derived] Pereira AJ, Moraes RB, Trott G, Santos MCD, Mocellin D, Andrade AYT, Miozzo AP, Paixao LCM, Schardosin RFC, Batista CL, Roldao ES, Silva CSM, Santos RDRMD, Cavalcanti MICES, Souza JMB, Matos LDNJ, Souza D, Neves JWC, Rech GS, Souza TMA, Silva GND, Itaqui CR, Yoshida SMS, Eid RAC, Camillis MLF, Genena KSR, Garcia LMC, Schaefer EC, Cidade PAP, Mariano NF, Sisto IR, Cruz ACLPD, Correa CL, Maia IR, Oliveira J, Carvalho A, Laguna MR, Ferraz LR, Teixeira C, Cavaliere YF, Zampieri FG, Rosa RG. The impact of a multicomponent telemedicine-based intervention on quality of life in adults with respiratory failure requiring mechanical ventilation: protocol for a cluster stepped-wedge randomized clinical trial (Tele-Rehab MV Trial). Crit Care Sci. 2025 Dec 15;37:e20250136. doi: 10.62675/2965-2774.20250136. eCollection 2025. PMID 41417397